CLINICAL TRIAL: NCT05059574
Title: The Effect of Breast Crawling After Vaginal Delivery on Breastfeeding Success and Mothers' Attitudes to Feeding Their Babies
Brief Title: Breast Crawling,Breastfeeding Success and Mothers' Attitudes to Feeding Their Babies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Dr. Kevser Ozdemir, PhD, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13092021
Record Dates: First submitted 2021-09-13; First posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Breast Feeding; Feeding Behavior
Keywords: Breast Crawling; Vaginal Delivery; Breastfeeding Success
MeSH Terms: conditions — Breast Feeding; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: While crawling to the breast is tried in the experimental group, biological breastfeeding will be applied in the control group.
Masking Description: Since there is no placebo group, masking will not be done.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Mothers in this group will begin their baby's first breastfeeding by crawling to the breast.
  Interventions: Behavioral: Breast Crawling
- Control group (No Intervention): Mothers in this group will begin their baby's first breastfeeding with biological breastfeeding.

INTERVENTIONS:
Behavioral: Breast Crawling — The mother's first breast-feeding of her baby is not routine biological breast-feeding, but as a cradle to the breast.
  Arms: Experimental group

SUMMARY:
It has been clearly demonstrated by the literature that the way of initiation of breastfeeding is highly correlated with the success and continuation of breastfeeding and the level of breastfeeding intention. Crawling to the breast is the reflex of seeking the breast by smelling the breastmilk of the newborn as the first form of breastfeeding. Although crawling to the breast is a studied subject in the international literature, it has remained only in the compilation stage in the national literature. The fact that research on breast crawling has not yet been conducted in our country constitutes the original value of this study. This study was planned to examine the effect of crawling to the breast after vaginal delivery compared to biological breastfeeding on breastfeeding success and mothers' attitude to feed their babies.

DETAILED DESCRIPTION:
Breastfeeding is one of the most effective ways to ensure child health and survival. Breast milk is the ideal food for babies. It is safe and clean. It contains antibodies that help protect against many common childhood diseases. Breast milk provides all the energy and nutrients a baby needs in the first months of life. However, about 2 out of 3 babies cannot be exclusively breastfed for the recommended 6 months.

WHO and UNICEF,

* early start of breastfeeding within 1 hour after birth,
* exclusive breastfeeding for the first 6 months of life
* Providing nutritionally sufficient and safe complementary (solid) foods in the 6th month, It recommends continuing breastfeeding up to 2 years of age. Early initiation of breastfeeding within 1 hour after birth protects the newborn from infection and reduces neonatal mortality. However, many infants and children do not receive optimal nutrition. For example, only about 44% of infants aged 0-6 months worldwide were exclusively breastfed during the 2015-2020 period.

Breastfeeding Success The most important reason for breastfeeding failure is the inability to start breastfeeding. For this reason, it is necessary to provide the necessary comfort of the mother in order to ensure breastfeeding success. In order to initiate and maintain a successful breastfeeding, mothers should be educated about being physically and mentally healthy, have a balanced diet, and be able to give breast milk with the right technique during pregnancy and the period following birth. Many mothers need help, especially when starting to breastfeed their first baby. A good start to breastfeeding affects the mother's determination to continue breastfeeding. However, difficulties encountered in breastfeeding during this period may lead to anxiety, causing mothers to lose their self-confidence and thus to a decrease in breastfeeding. Therefore, if the mother and baby are suitable, it is very important to initiate the first breastfeeding in this period called the 1st Stage (1st Reactive Period) after the birth.

Odent talked about the ability of a newborn to search for the breast for "that important first sucking action" within the first hour of opening his eyes to the world and to use the search reflex to find it. Widström et al. Crawling to the breast is defined as an organized, spontaneous behavior sequence of newborns to seek and move towards the nipple and initiate breastfeeding. In order to find the breast, newborns first use the stepping reflex to climb into the mother's belly, and then the search reflex to find the nipple, catch and suck. This is called newborn attachment or crawling to the breast. They stated that this behavior of the newborn can be observed in its most intact form within the first few hours of its birth.

The study was planned as a randomized controlled and experimental study in order to evaluate the effect of crawling on the breast after vaginal delivery on breastfeeding success and mothers' attitude to feed their babies.

Women who had vaginal delivery between October 2021 and April 2022 in the delivery room of S.B.Ü Darıca Farabi Training and Research Hospital will be included in the study.

The population of the research will be women who gave vaginal birth in the delivery room of S.B.Ü Darıca Farabi Training and Research Hospital between T October 2021 and April 2022, and the sample will be 68 women (34 control/34 experiment-intervention).

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the research,
* Vaginal birth,
* Over 18 years old,
* Able to read and write
* Can speak Turkish,
* Having a full-term and healthy birth (38-42 weeks old, born 2500-4000gr, born with a 5th minute apgar of 7 and above, no known congenital disease),
* Does not have a disease that prevents breastfeeding

Exclusion Criteria:

* Not voluntarily to participate in the research,
* Cesarean delivery,
* Having a health problem in which the mother or baby is at risk,
* Those who have a disease that prevents breastfeeding.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding success measurement | 2 years
  Determining the success of breastfeeding by getting a higher score on the LATCH Breastfeeding Diagnostic Scale in the experimental group, in which the first breast-feeding was applied by crawling to the breast compared to the control group.
Measuring mothers' feeding attitudes of their babies | 2 years
  In the experimental group in which the first breast-feeding was applied by crawling to the breast, the mothers' milk feeding behavior increased by getting a higher score on the "The Iowa Infant Feeding Attitude Scale" compared to the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The follow-up of the study data will be provided by both researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be kept by the researchers until the study is reported. After the study is published, it will contribute to the literature.
Access Criteria: After the study is reported and published, it will be shared.

REFERENCES:
- [Background] Hym C, Forma V, Anderson DI, Provasi J, Granjon L, Huet V, Carpe E, Teulier C, Durand K, Schaal B, Barbu-Roth M. Newborn crawling and rooting in response to maternal breast odor. Dev Sci. 2021 May;24(3):e13061. doi: 10.1111/desc.13061. Epub 2020 Dec 5. PMID 33174352
- [Background] Henderson A. Understanding the breast crawl: implications for nursing practice. Nurs Womens Health. 2011 Aug-Sep;15(4):296-307. doi: 10.1111/j.1751-486X.2011.01650.x. No abstract available. PMID 21884495
- [Background] Heidarzadeh M, Hakimi S, Habibelahi A, Mohammadi M, Shahrak SP. Comparison of Breast Crawl Between Infants Delivered by Vaginal Delivery and Cesarean Section. Breastfeed Med. 2016 Aug;11(6):305-308. doi: 10.1089/bfm.2015.0168. Epub 2016 May 12. PMID 27171469